CLINICAL TRIAL: NCT05427448
Title: Clinical Validation of the Use of Blood Biomarkers for the Diagnosis and Monitoring of Alzheimer's Disease
Brief Title: Validation of Blood Biomarkers for Alzheimer's Disease
Acronym: ALZAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL21_0586
Record Dates: First submitted 2022-06-17; First posted 2022-06-22 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Dementia; Tauopathies
Keywords: blood; Alzheimer; biomarker
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia; Tauopathies

STUDY DESIGN:
Intervention Model Description: Prospective consecutive enrollment clinical trial to assess the diagnostic performance (sensitivity, specificity) of blood biomarkers for Alzheimer's disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective multisite clinical trial with consecutive recruitment. (Experimental): Patients consulting in memory clinics from Montpellier, Nîmes, or Perpignan. CSF AD biomarkers performed for diagnostic purpose in clinical routine practice
  Interventions: Diagnostic Test: Measurement of amyloid and pTau blood biomarkers

INTERVENTIONS:
Diagnostic Test: Measurement of amyloid and pTau blood biomarkers — Detection of plasma Amyloid beta 1-40 and 1-42 peptide and phosphorylated tau isoforms.

SUMMARY:
Alzheimer's disease (AD) has gradually become one of the major global public health issues due to its prevalence, which increases with age and life expectancy, and the economic cost of caring for patients whose cognitive decline progressively leads to loss of functional autonomy.

The diagnosis of AD is based on a multidisciplinary approach, involving, among other things, evaluation of the medical history together with clinical symptoms and signs, neuropsychological tests and neuroimaging. The quantification of cerebrospinal fluid (CSF) core biomarkers (amyloid beta peptides [Ab1-40 and Ab1-42], total tau [t-tau] and its phosphorylated form on threonine 181 [p-tau(181)]) has progressively proven utility for the diagnosis of AD and its prodromal forms. CSF biomarkers are now included in international guidelines for the diagnosis of AD in research settings and clinical practice and the Alzheimer's Association appropriate use criteria for the use of lumbar puncture and CSF testing in the diagnosis of AD have been published. Such biochemical diagnostics are currently implemented in many specialized centers around the world.

Recent progress in the biological diagnosis of AD is considerable, with the possibility, thanks to ultra-sensitive tests realized notably with the SIMOA technology, of having Ab1-40, Ab1-42, t-tau and p-tau(181) also detectable in the blood using commercial kits. The performance for AD detection has been evaluated by many groups including on retrospective samples.

It is now essential to evaluate the interest of blood-based biomarkers of AD, prospectively and in real life condition to confront them with pre-analytical and analytical variabilities. It is also important to position them in relation to CSF analysis and AD management, from risk assessment, diagnosis, to therapeutic strategies.

DETAILED DESCRIPTION:
Rationale of the project:

Recent progress in the biological diagnosis of Alzheimer's disease (AD) is considerable, with the possibility, thanks in particular to ultra-sensitive tests, of having relevant blood biomarkers. These biomarkers, mainly represented by amyloid peptides, tau proteins and neurofilaments, make it possible to consider a stratification of patients according to different classifications, including the ATN scale. Their diagnostic value has been mainly tested on retrospective samples and it is now essential to use them prospectively to confront them with pre-analytical and analytical variability. It is also important to position them in relation to CSF analysis and AD management, from risk assessment, diagnosis, to therapeutic strategies.

Main objective:

To evaluate, in a prospective consecutive enrollment clinical trial, the diagnostic performance (sensitivity, specificity) of blood biomarkers for Alzheimer's disease.

Secondary objectives:

* Interest of blood biomarkers for detection of normal/pathological CSF profiles.
* Interest of blood biomarkers for other disease including, amyloid angiopathy, frontotemporal dementia (FTD) or lewy body disease (LBD).

Methodology:

The investigator's laboratory daily receives CSF samples from regional "memory clinics" (mainly from Montpellier, Nîmes, Perpignan) for Aß40, Aß42, t-Tau and p-Tau(181) assays. The results of these tests performed weekly on an automated platform are used by neurologists for the diagnosis of AD. In this non-interventional multi-center clinical trial, with the informed consent of patients, one tube of plasma in addition to CSF is collected. In parallel with the CSF, amyloid peptides and plasma p-Tau is measured. The ApoE4 status will also be determined using MS as previously published by the investigator's group. Plasma biomarkers will then be combined to confirm the presence of AD, as has already been done on retrospective samples by the investigator's laboratory and others. Considering a disease prevalence rate of 20% in the screened population, and to reach a sensitivity of 80% and a specificity close to 90%, it is necessary to include a total of 311 patients in order to obtain an estimate of sensitivity and specificity with a 95% accuracy of +/- 10%. The lost to follow-up rate of about 10% requires the enrollment of 342 patients. The diagnostic performance of this profile will be compared to that of CSF, as well as to the diagnosis assessed by a multidisciplinary team one year after sampling.

Expected benefit:

The confirmation that blood biomarkers of AD achieve satisfactory diagnostic performance in a clinical setting allows them to be considered in routine use, as a less invasive method, thus with greater acceptance and also the possibility of longitudinal use. The benefit also lies in the evaluation of the interest of supplemental biomarkers such as NfL, for related diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients consulting in memory clinics from Montpellier, Nîmes, or Perpignan.
* Age >= 18 years old
* CSF AD biomarkers performed for diagnostic purpose in clinical routine practice
* Having given their written and enlightened consent
* Affiliated or beneficiary of the national health insurance

Exclusion Criteria:

* Contraindication or refusal of lumbar puncture
* Patient deprived of freedom, by court or administrative order, or major protected by law
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of blood biomarkers for Alzheimer's disease | 24 months
  Calculate the performance (sensitivity, specificity) of biomarkers, alone or in combination, for the detection of Alzheimer's disease as defined by the McKhann criteria.

SECONDARY OUTCOMES:
Prediction of CSF profile | 24 months
  Calculate the performance (sensitivity, specificity) of biomarkers, alone or in combination, for the detection of normal vs pathological CSF profile (ATN)
Diagnostic performance of blood biomarkers for FTD or LBD | 24 months
  Calculate the performance (sensitivity, specificity) of biomarkers, alone or in combination.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Lehmann, MD PhD, Principal Investigator — University Hospital, Montpellier
Locations (3):
- France (3):
  - Montpellier University Hospital, Montpellier, Occitanie
  - Nîmes University Hospital, Nîmes, Occitanie
  - Perpignan Regional Hospital, Perpignan, Occitanie

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Delaby C, Alcolea D, Hirtz C, Vialaret J, Kindermans J, Morichon L, Fortea J, Belbin O, Gabelle A, Blennow K, Zetterberg H, Lleo A, Lehmann S. Blood amyloid and tau biomarkers as predictors of cerebrospinal fluid profiles. J Neural Transm (Vienna). 2022 Feb;129(2):231-237. doi: 10.1007/s00702-022-02474-9. Epub 2022 Feb 15. PMID 35169889
- [Result] Lleo A, Zetterberg H, Pegueroles J, Karikari TK, Carmona-Iragui M, Ashton NJ, Montal V, Barroeta I, Lantero-Rodriguez J, Videla L, Altuna M, Benejam B, Fernandez S, Valldeneu S, Garzon D, Bejanin A, Iulita MF, Camacho V, Medrano-Martorell S, Belbin O, Clarimon J, Lehmann S, Alcolea D, Blesa R, Blennow K, Fortea J. Phosphorylated tau181 in plasma as a potential biomarker for Alzheimer's disease in adults with Down syndrome. Nat Commun. 2021 Jul 14;12(1):4304. doi: 10.1038/s41467-021-24319-x. PMID 34262030
- [Result] Alcolea D, Delaby C, Munoz L, Torres S, Estelles T, Zhu N, Barroeta I, Carmona-Iragui M, Illan-Gala I, Santos-Santos MA, Altuna M, Sala I, Sanchez-Saudinos MB, Videla L, Valldeneu S, Subirana A, Pegueroles J, Hirtz C, Vialaret J, Lehmann S, Karikari TK, Ashton NJ, Blennow K, Zetterberg H, Belbin O, Blesa R, Clarimon J, Fortea J, Lleo A. Use of plasma biomarkers for AT(N) classification of neurodegenerative dementias. J Neurol Neurosurg Psychiatry. 2021 Nov;92(11):1206-1214. doi: 10.1136/jnnp-2021-326603. Epub 2021 Jun 8. PMID 34103344
- See also: Clinical proteomics — https://www.chu-montpellier.fr/fr/irmb/laboratoires-et-plateformes-hospitalieres